CLINICAL TRIAL: NCT06548477
Title: Effectiveness of Human Albumin for Clinical Outcome in Aneurysmal Subarachnoid Hemorrhages: A Protocol for Randomized Controlled (Hash) Trial.
Brief Title: Human Albumin for Clinical Outcome in Aneurysmal Subarachnoid Hemorrhages
Acronym: HASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr Arshad Ali, Consultant neurosurgery, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MR-01-24-229
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: HASH trial, Human Albumin, Subarachnoid hemorrhage, Aneurysmal, Effectiveness, Clinical Outcome, Protocol
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Albumin group) (Experimental): Intervention group will receive of intermittent boluses of human albumin plus standard fluid therapy (with crystalloids only) to maintain a euvolemic fluid balance.
  Interventions: Drug: Human albumin
- Control (crystalloid group) (No Intervention): Control group will receive only standard fluid therapy with crystalloid solutions with intermittent boluses crystalloid solution to maintain euvolemic balance

INTERVENTIONS:
Drug: Human albumin — Patients in intervention arm will also receive intermittent boluses of 20 percent human albumin (in addition to standard fluid therapy) that will be administered with dosage regimen of 1.25gm/kg of body weight per 24 hours. The maximum total calculated dose/volume of albumin for the patient will be infused @ 34 ml/hour (over 3 hours) and will be divided in 3 boluses, spaced at 8 hours intervals. During intervention period, duration of treatment (7-day study period) will cover the peak period of cerebral vasospasm from day 4th until 10th day. Albumin administration will be tailored according to the targeted values set for euvolemic fluid balance in each patient. Before randomization (within 72 hours post-ictus) and after day-10 (from day 11th-14th, patient will only receive standard fluid therapy.
  Arms: Intervention group (Albumin group)

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is a dreadful acute neurological condition with overwhelmingly high rate of associated morbidities and mortality. Despite leaping advancement in neurosurgical techniques and imaging modalities, there is no substantiative improvement in overall prognosis for aSAH. Cerebral vasospasm remains the predominant cause of associated morbidities. Human albumin has been used in different neurological conditions including head trauma, intracerebral hemorrhages, and ischemic strokes with favorable outcome. However, its beneficial use in aSAH has not been sufficiently explored until recently a published systematic review by our team. In view of scarcity of published data and lack of robust evidence, our group has designed for the first ever RCT to compare the use human albumin-enhanced fluid management versus standard fluid therapy with crystalloids in patients with aSAH.

This single center open label, prospective, parallel group randomized control trial will be conducted at Hamad General Hospital, Doha-Qatar from August 2024 to July 2027. A sample size of 84 (42 in each arm) has been calculated to detect as sufficient to detect a clinically significant difference in modified Rankin Scale good score between two groups (human-albumin induced volume expansion therapy versus crystalloid only) for fluid management in aneurysmal subarachnoid hemorrhages patients. Primary outcome will be based on dichotomized modified Rankin scale [(Good grades (0-2) and poor grades (3-6)], while secondary outcome will include symptomatic vasospasm, transcranial doppler velocities, and Pulse Index Contour Cardiac Output (PiCCO) parameters.

The trial aims to provide firsthand evidence on the beneficial use of human albumin to achieve optimal fluid management regime to explore its potential role to improve clinical outcome in patients with aSAH.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a fatal neurosurgical emergency that may reach to a mortality of up to nearly 60% within one month of symptoms onset in untreated cases. Accounting for almost 5% of all stroke cases, aSAH predominantly affects the working age population with significant socioeconomic effect due to its impact on their quality of healthy life. Despite refined contemporary neurosurgical techniques and advancements in neurocritical care, secondary/delayed ischemia neurological deficits due to cerebral vasospasm, have been implicated as the main contributing factor, related to poor clinical outcome in nearly 30% of the patients. Although, over the years, many different treatment modalities have been used to counter the detrimental effects of vasospasm including calcium channel blockers and triple-H therapy (hypervolemic, hemodilution, hypertension) with no substantiative improvement in clinical outcome and a search for an effective management strategy continues.

In aSAH, hyponatremia due to increased release of natriuretic factors and reduction in intravascular volume have been attributed to cause clinical vasospasm and delayed ischemic neurological deficits as a part of natural course of the disease. Reduced cerebral blood flow during aSAH has been explained based on two etiological factors. Firstly, immediately with the clinical onset of aSAH, there is a generalized decrease in brain oxidative metabolism that contributes to drop in global cerebral blood flow (CBF). This disruption in brain metabolic harmony is primarily caused by presence of toxic blood products in subarachnoid spaces although other contributing factors including acute hydrocephalus, brain edema and rise in intracranial pressure may also play their roles to already compromised CBF. Secondly, during the course of subsequent days to weeks when cerebral vasospasm sets in, it can further cause drop in CBF and cerebral metabolism. This drop in CBF is topographically heterogenous in brain parenchyma and this manifests as the delayed cerebral ischemia causing neurological deficits. Based on these pathophysiological mechanisms, the standard use of hypervolemic therapy was rationalized in neurosurgical practice in the past to mitigate the detrimental effects of hypoperfusion and it used to be achieved by routine use of crystalloids/isotonic solutions and complementary colloidal agents including dextran, hypertonic saline and human albumin in neurocritical care.

In animal studies with rat models for acute focal ischemia, albumin treatment has effectively reduced size of penumbra. In contemporary clinical practice, the beneficial effects of human albumin has been investigated in cerebral strokes, acute brain injury, intracranial hemorrhages, including aSAH with promising results. In a pilot study conducted by Suarez et al (ALISAH) for a clinically safe dosage regimen for aSAH, it has also been observed that the use of albumin may be effective to prevent the deleterious effects of cerebral vasospasm by enhanced CBF leading to improvements in neurological outcome in aSAH patients. Ali A. et al recently published a systematic review that underscores obvious gaps in literature for the use of human albumin with no randomized control trial published to-date and highlighting the lack of any robust clinical evidence for the role of albumin to treat cerebral vasospasm in aSAH This single center RCT will aim to explore potential beneficial role of human albumin to improve clinical outcome in patients with aSAH.

ELIGIBILITY:
Inclusion criteria

* Age limits of participants will be between 18 and 80 years with either gender (male or female).
* Clinical presentation with the first of symptom of aSAH must be within 72 hours before randomization.
* Clinical manifestation must be suggestive of aSAH that may include classical thunderclap headache, cranial nerve deficits, changes in level of consciousness, neck rigidity and neurological deficits.
* All cases with WFNS grade 1 to 5 (at the time of randomization) will be recruited in the study.
* Head computed tomography demonstrates evidence of SAH (graded on Claassen's scale).
* Diagnostic cerebral angiography shows a saccular aneurysm/s, consistent with clinical presentation of SAH.
* Definitive treatment of ruptured aneurysm/s (with clipping or coiling of combined) must be carried out within 72 hours prior to randomization.
* An informed consent by patient or surrogate representative, must be duly signed and dated.

Exclusion criteria

* Timing of first symptom of SAH cannot be reliably ascertained.
* Cerebral angiogram negative SAH.
* Cerebral angiography showing mycotic/traumatic/fusiform aneurysm/s.
* Symptomatic vasospasm or angiographic (on TCD or CTA) sets in before recruitment within 72 hours.
* History of clinical findings/hospitalization due to heart failure within the past 6 months,
* Albumin administration prior to randomization in the same hospital admission.
* History of acute myocardial infarction (MI) within past 3 months.
* Any clinical presentations or electrocardiography (ECG) findings suggestive of acute MI on current admission.
* ECG evidence and/or clinical findings of 2nd or 3rd degree heart block or arrhythmias causing hemodynamic changes.
* Echocardiogram done before intervention/randomization showing an ejection fraction of <40%.
* A creatinine level of >2.0 mg/dl or a creatinine clearance of <50 ml/min
* Pregnancy, lactation, or parturition within previous 30 days
* Any allergies to any ingredient in human albumin preparation.
* A prior severe physical disability (mRS >2) that may hamper assessment of clinical outcome.
* Advanced chronic obstructive pulmonary diseases (with FEV1 <50%) may manifest as frequent episodes significantly affecting the overall quality of life.
* Hepatic failure or suspected liver dysfunction due to deranged liver functions, decreased serum albumin levels, high bilirubin levels with/without peripheral edema and hepatic encephalopathy.
* Patient has been already enrolled in another study involving a drug administration.
* Patient suffering from terminal diseases with life expectancy < 6 months
* If patient speaks any other language in which consent has not been translated.
* In case, patient drops out/withdraws from study or transferred out of state of Qatar and therefore lost to follow up short of 3-month follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Dichomatized modified Rankin Scale (mRS) | Endpoints for primary outcome measures (values of mRS) will be assessed on Day-14 and at 3 month follow up.
  Primary clinical outcome will be based on dichotomized modified Rankin Scale [(Good grades (0 -2) and poor grades (3-6)]. Primary outcome measures (values of mRS) will be compared between study arms to assess difference in the effect size of the intervention.

SECONDARY OUTCOMES:
Development of Symptomatic vasospasm (with/without new onset infarctions on unenhanced Computed Tomography scan, transcranial doppler velocities (daily average) and PiCCO parameters (daily average values) | Endpoint for secondary outcome is at day-14.
  Secondary outcomes will include symptomatic vasospasm (with/without new onset infarctions on unenhanced Computed Tomography scan), transcranial doppler velocities (daily values), and all Pulse index Contour Cardiac Output (PiCCO) parameters (daily average values). On 14th day endpoint, a mean of all cumulative daily averaged values will be recorded for secondary outcome measures for; 1) the study period (4th-10th day) and 2) subsequently without albumin therapy (from day 11th -14th day) on Day-14 end-point. These secondary outcome measures will be compared between study arms to assess difference in the effect size of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Ali, MBBS, MPH, FCPS, MSc, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

REFERENCES:
- [Background] Ali A, Rajeswaran AB, Shaikh N, Al-Rumaihi G, Al-Sulaiti G. Role of albumin-induced volume expansion therapy for cerebral vasospasm in aneurysmal subarachnoid hemorrhage: A systematic review. J Neurosci Rural Pract. 2023 Oct-Dec;14(4):582-590. doi: 10.25259/JNRP_372_2023. Epub 2023 Oct 3. PMID 38059246
- [Background] Suarez JI, Shannon L, Zaidat OO, Suri MF, Singh G, Lynch G, Selman WR. Effect of human albumin administration on clinical outcome and hospital cost in patients with subarachnoid hemorrhage. J Neurosurg. 2004 Apr;100(4):585-90. doi: 10.3171/jns.2004.100.4.0585. PMID 15070109
- [Derived] Ali A, Khan M, Shaikh N, Mohamad AE, Al-Maadhadi M, Shah N, Al-Najjar Y, Salam A, Al-Rumaihi G, Ayyad A, Belkhair S, Al-Sulaiti G. Effectiveness of human albumin for clinical outcome in aneurysmal subarachnoid hemorrhages: a protocol for randomized controlled (HASH) trial. Trials. 2025 Feb 14;26(1):53. doi: 10.1186/s13063-025-08762-5. PMID 39953562